CLINICAL TRIAL: NCT00292461
Title: A Study for Evaluating the Efficacy and Safety of Zonisamide and Lamotrigine (Lamictal) for Subjects With Refractory Simple Partial, Complex Partial or Partial With Secondary Generalized Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2090-AS886-202
Record Dates: First submitted 2006-02-14; First posted 2006-02-16 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2009-08

CONDITIONS: Epilepsy
Keywords: Epilepsy; seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Zonisamide; Lamotrigine

ARMS (2):
- zonisamide (Active Comparator): tablet
  Interventions: Drug: Zonisamide
- lamotrigine (Active Comparator): tablet
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Zonisamide — Tablet once or twice daily orally for 16 weeks
  Arms: zonisamide
Drug: Lamotrigine — Tablet once daily orally for 16 weeks
  Arms: lamotrigine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of zonisamide for anti-epilepsy drugs (AEDs) treated subjects with refractory simple partial, complex partial or partial with secondary generalized seizures.

ELIGIBILITY:
Inclusion criteria:

* Subjects must sign and date the informed consent form
* Clinical diagnosis as refractory epilepsy

Exclusion criteria:

* Progressive neurologic disease
* Serious psychiatric disease
* Hemolytic anemia
* G6PD (glucose-6-phosphate dehydrogenase) deficiency
* Acute intermittent porphyrias
* Subjects who have received study drugs (Zonisamide, Lamotrigine) in the past
* Drug or alcohol addiction
* Renal impairment (serum creatinine ≧ 1.5 mg/dl), or hepatic abnormality (ALT or AST > 2x ULN)
* Stevens-Johnson syndrome
* Progressive exfoliative dermatitis
* Pregnant, lactating or of childbearing potential female
* Regularly taking oral contraceptives
* Hypersensitivity to study drugs
* Severe cardiac disease (New York Heart Association Functional Class III and IV)
* History of malignancy within 5 years

  * Taking valproic acid within 7 days prior to screening
  * Subjects with simple partial seizures without motor component

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-03; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Hui Cheng, Study Director — Eisai Taiwan
Locations (8):
- China (8):
  - Changhua Christian Hospital, Changhua, Taiwan
  - Chang-Gung Memorial Hospital (CGMH), Kaohsiung, Taiwan
  - Chang-Gung Memorial Hospital (CGMH), Linkou, Taiwan
  - China Medical University Hospital (CMUH), Taichun, Taiwan
  - National Cheng Kung University Hospital, Tainan, Taiwan
  - Chang-Gung Memorial Hospital (CGMH), Taipei, Taiwan
  - Taipei Tzu Chi General Hospital, Taipei, Taiwan
  - Taipei Veterans General Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Zonegran: once or twice daily orally for 16 weeks
- Lamotrigine: once daily orally for 16 weeks
Period: Overall Study
Arm/Group | Zonegran | Lamotrigine
Started | 34 | 30
Completed | 24 | 24
Not Completed | 10 | 6
Not completed — Adverse Event | 4 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 4 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonegran | Lamotrigine | Total
Number analyzed (Participants) | 34 | 30 | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 38.3 (11.5) | 35.0 (9.8) | 36.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 18 | 13 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 34 | 30 | 64
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 34 | 30 | 64

OUTCOME MEASURES:

1. Primary Outcome: The Percentage Change of Monthly Seizure Frequency at the End of the 16-week Treatment From Baseline
Description: Percentage Change of Frequency = (T-B)/B*100% T= Total seizure frequency during maintenance dose period / maintenance dose period (weeks)* 4 B= The monthly seizure frequence with one month prior to enrollment
Time Frame: Baseline and 16 weeks
Population: ITT (intent-to-treat)
Measure: Median (Full Range); unit: percent change
Arm/Group | Zonegran | Lamotrigine
Number analyzed (Participants) | 24 | 24
percent change | -32.7 [-100 to 180.0] | -35.6 [-100 to 444.4]
Statistical Analysis 1: Comparison: Zonegran vs Lamotrigine; Test type: Superiority or Other; p = 0.240, ANOVA

2. Secondary Outcome: Global Assessment of Efficacy by Physician at the End of 16-week Treatment Period
Time Frame: Baseline and 16 weeks
Measure: Number; unit: participants
Arm/Group | Zonegran | Lamotrigine
Number analyzed (Participants) | 24 | 24
participants
  Greatly improved | 5 | 4
  Somewhat improved | 9 | 15
  No change | 10 | 5
  Somewhat worsened | 0 | 0
  Greatly worsened | 0 | 0
Statistical Analysis 1: Comparison: Zonegran vs Lamotrigine; Test type: Superiority or Other; p = 0.460, Cochran-Mantel-Haenszel

3. Secondary Outcome: Global Assessment of Efficacy by Participants at the End of the 16-week Treatment Period
Time Frame: Baseline and 16 weeks
Measure: Number; unit: participants
Arm/Group | Zonegran | Lamotrigine
Number analyzed (Participants) | 24 | 24
participants
  Greatly improved | 3 | 8
  Somewhat improved | 14 | 12
  No change | 4 | 4
  Somewhat worsened | 3 | 0
  Greatly worsened | 0 | 0
Statistical Analysis 1: Comparison: Zonegran vs Lamotrigine; Test type: Superiority or Other; p = 0.079, Cochran-Mantel-Haenszel

4. Secondary Outcome: Response Rate: Defined as the Percentage of Participants With >= 50% Reduction of Monthly Seizure Frequency at the End of 16-week Treatment From Baseline.
Time Frame: Baseline and 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Zonegran | Lamotrigine
Number analyzed (Participants) | 24 | 24
percentage of participants | 45.8 | 45.8
Statistical Analysis 1: Comparison: Zonegran vs Lamotrigine; Test type: Superiority or Other; p = 0.860, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Arm/Group | Zonegran | Lamotrigine
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/30
Other Adverse Events (participants affected / at risk) | 20/34 | 20/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zonegran (N=34) | Lamotrigine (N=30)
Lumber contusion (Musculoskeletal and connective tissue disorders) | 0 | 1
nystagmus (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zonegran (N=34) | Lamotrigine (N=30)
Disturbance in attention (Nervous system disorders) | 1 | 0 — Derived from Table for all drug-related AEs
dizziness (Nervous system disorders) | 2 | 2 — Derived from Table for all drug-related AEs
Gait disturbance (Nervous system disorders) | 0 | 1 — Derived from Table for all drug-related AEs
insomnia (Nervous system disorders) | 0 | 2 — Derived from Table for all drug-related AEs
nystagmus (Nervous system disorders) | 0 | 1 — Derived from Table for all drug-related AEs
somnolence (Nervous system disorders) | 2 | 2 — derived from Table for all drug-related AEs
White blood cell urine positive (Investigations) | 1 | 0 — Derived from Table for all drug-related AEs
Blood alkaline phosphatase increased (Investigations) | 2 | 0 — Derived from Table for all drug-related AEs
Electrocardiogram abnormal (Investigations) | 1 | 0 — Derived from Table for all drug-related AEs
Hepatic enzyme abnormal (Investigations) | 3 | 0 — Derived from Table for all drug-related AEs
Red blood cell urine positive (Investigations) | 2 | 0 — Derived from Table for all drug-related AEs
Weight decreased (Investigations) | 1 | 0 — Derived from Table for all drug-related AEs
Mood altered (Psychiatric disorders) | 0 | 1 — Derived from Table for all drug-related AEs
nausia (Gastrointestinal disorders) | 0 | 1 — Derived from Table for all drug-related AEs
Abdominal distention (Gastrointestinal disorders) | 0 | 1 — Derived from Table for all drug-related AEs
anorexia (Metabolism and nutrition disorders) | 1 | 1 — Derived from Table for all drug-related AEs
malaise (General disorders) | 1 | 0 — Derived from Table for all drug-related AEs
splenomegaly (Blood and lymphatic system disorders) | 1 | 0 — Derived from Table for all drug-related AEs
Hepatic function disorders (Hepatobiliary disorders) | 1 | 0 — Derived from Table for all drug-related AEs
contusion (Musculoskeletal and connective tissue disorders) | 0 | 1 — Derived from Table for all drug-related AEs
pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 — Derived from Table for all drug-related AEs
rash (Skin and subcutaneous tissue disorders) | 1 | 2 — Derived from Table for all drug-related AEs
diplopia (Eye disorders) | 0 | 3 — Derived from Table for all drug-related AEs
Vision blurred (Eye disorders) | 0 | 1 — Derived from Table for all drug-related AEs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No